CLINICAL TRIAL: NCT06685822
Title: Expanding Autism Diagnostic Biomarkers to Kenya
Acronym: KinleyET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Rebecca McNally Keehn, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23559
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Children participate in eye-tracking activity (Experimental): Children enrolled in the HEAL-R Autism at MTRH study will be enrolled into the study. Research participation includes a one-time eye-tracking activity in which the child will view a series of different pictures and movies while their eye movements and pupil diameter are tracked and recorded.
  Interventions: Diagnostic Test: Eyelink Portable Duo

INTERVENTIONS:
Diagnostic Test: Eyelink Portable Duo — Eye-tracking data will be collected using a commercially-available remote eye-tracking system (Eyelink Portable Duo). Eye movements and pupil diameter will be collected while participants view a series of developmentally appropriate pictures and movies. The eye-tracker consists of two cameras; one that monitors eye movements and a second scene camera that monitors head movements, which permits eye tracking to take place without any equipment touching the child. Children will be asked to sit in highchair or on their the lap of the caregiver and will face a computer monitor. After a sticker is applied to the forehead of the child and brief eye-movement calibration completed, next visual stimuli (i.e., pictures and videos) will be presented on a laptop computer monitor that is placed at approximately 60-80cm from the child. The eye tracking portion of the visit will last approximately 15 minutes or until the child is no longer able to attend to pictures/videos.

SUMMARY:
The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series of eye-tracking measures.

DETAILED DESCRIPTION:
The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series (less than 15 mins) of eye-tracking measures (e.g., looking time, pupil diameter, oculomotor dynamics), which may be associated with autism in young children. The investigators will recruit children from Moi Teaching and Referral Hospital (MTRH; Eldoret, Kenya) previously enrolled in the Health Equity Advancing through Learning Health Systems Research (HEAL-R) Autism at MTRH study (IREC/664/2023, approval number 0004633)

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the HEAL-R Autism at MTRH study
* Children ages 14-72 months
* Caregivers of children must speak Kiswahili (local language) or English.

Exclusion Criteria:

* Children not enrolled in the HEAL-R Autism at MTRH study
* Children younger than 14 months or older than 72 months
* Caregivers of children do not speak Kiswahili (local language) or English.

Ages: 14 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Agreement between eye-tracking biomarker score and autism diagnosis | Day 1
  Group (autism presence/absence) differences in the composite eye-tracking biomarker score, a consolidated measure based on eye-tracking indices, will be tested to determine whether this metric is predictive of autism diagnosis. Clinical diagnosis was obtained based upon a standardized clinical evaluation in the parent study. The evaluation included: 1) a semi-structured caregiver(s) clinical interview to gather information about developmental history and autism symptoms and 2) a battery of standardized child clinical observational measures. Eye-tracking biomarkers will be recorded during a brief one-time research visit.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Keehn, PhD, Principal Investigator — Purdue University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No